CLINICAL TRIAL: NCT03674268
Title: Psychometric Properties of the Spanish Version of the Contraversive Pushing Scale
Brief Title: Psycometric Properties of Pushing Scale
Status: Completed | Type: Observational
Sponsor: Guadarrama Hospital (Other)
Collaborators: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Other Study IDs: 4.0
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-10

CONDITIONS: Balance; Functionality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Management of the Contraversive Pushing Scale — Scale of evaluation of trunk control and pushing behavior in patients with stroke.

SUMMARY:
Psycometric properties of a scale

DETAILED DESCRIPTION:
After a period of training in the administration of the CPS, a pilot will be conducted with 10 patients who meet the inclusion-exclusion criteria and after signing the informed consent document, in which the 4 researchers will administer the CPS during two sessions on consecutive days, with the objective of evaluating the test-retest and intra-observer reliability, minimize the differences of criteria in its application and, if necessary, write an instruction manual.

Once each patient has signed the informed consent document and it has been verified that the inclusion criteria are met, it will be assigned an Identification Number (ID) that will relate it to your Medical Record (IDHC) by simple coding; The custody of the file with the relation of each ID with its HC will be borne by the principal investigator. Likewise, each observer will be assigned an identification number in order to blind the researcher who performs the statistical analysis. The patients included in the study will be evaluated, through the Spanish version of the CPS, by two of the researchers with an interval of 10 minutes between each evaluation, repeating this same procedure the next day. These evaluation sessions will be carried out throughout the treatment period, repeating on days 1, 15 and 28 of the period of admission of the included patients. Two researchers will evaluate the patients treated in the morning shift and the other two those treated in the afternoon shift of the Physiotherapy Service of the Guadarrama Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign the corresponding informed consents and information sheet before any evaluation / procedure related to the study is conducted.
* Male or female, ≥18 years of age at the time of consent.
* Have the diagnosis of ischemic or hemorrhagic hemispheric stroke without excluding other causes (surgery, cancer, etc ...).
* Enter for the first time in the Guadarrama Hospital to receive physiotherapy treatment.

Exclusion Criteria:

* A patient can not be recruited in this study if they have severe cognitive impairment, moderate-severe language problems, or severe vision or hearing deficits that prevent compression and active collaboration during evaluation tests.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of stroke who enter the Guadarrama Hospital, meet the inclusion / exclusion criteria and agree to participate in the study after signing the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Contraversive Pushing Scale score | 4 weeks
  Scale of evaluation of trunk control and pushing behavior in patients with stroke.

CONTACTS AND LOCATIONS:
Overall Officials: J.Nicolas Cuenca Zaldivar, Principal Investigator — Guadarrama Hospital
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The statistical analysis plan and the analytical code will be available in .html and .rmd format as well as the file with the raw data.
Supporting Information: Analytic Code
Time Frame: The data will be available permanently once the statistical analysis is complete.
Access Criteria: The data will be available freely and publicly.